CLINICAL TRIAL: NCT02133885
Title: Angiotensin and Neuroimmune Activation in Hypertension
Brief Title: Study 2: Effect of Minocycline Treatment on Drug-Resistant Hypertensive Patients
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: This study was never started and no participants were enrolled.
Sponsor: University of Florida (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB201500594-N; RO1HL3361028 (Other: National Heart, Lung, and Blood Institute (NHLBI)); 2013-00102 Study 2 (Other: University of Florida); R01HL132448-01 (NIH)
Record Dates: First submitted 2014-05-06; First posted 2014-05-08 (Estimated); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Hypertension
Keywords: Resistent Hypertension; Systolic Blood Pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Minocycline Group (Active Comparator): These subjects will start with minocycline for 16 weeks, followed by a washout period for 3 weeks, then will receive a placebo for 16 weeks, followed by a washout period for 3 weeks, then will finish with minocycline for 16 weeks.
  Interventions: Drug: Minocycline Group
- Placebo Group (Placebo Comparator): These subjects will start with placebo (this will look like minocycline) for 16 weeks, followed by a washout period for 3 weeks, then will receive a minocycline for 16 weeks, followed by a washout period for 3 weeks, then will finish with placebo for 16 weeks.
  Interventions: Other: Placebo Group

INTERVENTIONS:
Drug: Minocycline Group — These subjects will start with minocycline for 16 weeks, followed by a washout period for 3 weeks, then will receive a placebo for 16 weeks, followed by a washout period for 3 weeks, then will finish with minocycline for 16 weeks.
  Arms: Minocycline Group
Other: Placebo Group — These subjects will start with placebo (tablet looking just like minocycline) for 16 weeks, followed by a washout period for 3 weeks, then will receive minocycline for 16 weeks, followed by a washout period for 3 weeks, then will finish with placebo for 16 weeks.
  Arms: Placebo Group

SUMMARY:
Hypertension (HTN) is the single most prevalent risk factor for cardiovascular disease, diabetes, obesity and metabolic syndrome. Despite advances in life style modification and multi-drug therapies, 20-30% of all hypertensive patients remain resistant.

These individuals exhibit autonomic dysregulation due to elevated sympathetic activity and norepinephrine spillover, and low parasympathetic activity. It is generally accepted that this uncontrolled, resistant HTN is primarily "neurogenic" in origin, involving over activity of the sympathetic nervous system that initiates and sustains HTN. Thus, a mechanism-based breakthrough is imperative to develop novel strategies to prevent and perhaps eventually cure neurogenic hypertension (NH).

This study is a double-blind, placebo-controlled, cross-over design to test the hypothesis that minocycline treatment would produce antihypertensive effects in drug-resistant neurogenic hypertensive individuals.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, cross over design to evaluate the effects of minocycline in patients with resistent hypertension. After providing informed consent, patients will have baseline and followup visits during which a brief physical examination will be performed, medical history, assessment of medication compliance and tolerance, and vital signs will be completed.

Subjects will undergo blood (lipid panel, high sensitivity-C reactive protein, high sensitivity troponin, glucose, metabolic profile, lipid panel, Cystatin C and albumin) and urine studies at the baseline visit and at 16, 19, 35 and 54 weeks. Patients will have ambulatory BP monitoring at baseline and at the end of each treatment period.

Patients will be randomized to drug scheme A or B. One scheme will follow the following order: 16 weeks of minocycline, followed by a 3 week wash out period, then 16 weeks of placebo, then 3 weeks of wash out and a final 16 week period of minocycline. The other scheme will consist of 16 weeks of placebo, followed by 3 week wash out period, followed by 16 weeks of minocycline, then 3 week wash out and a final 16 weeks of placebo. Study visits will occur at study entry (baseline/randomization), 16 weeks, 19 weeks, 35 weeks, 38 weeks, and 54 weeks for each group. Patient participation will end after 56 weeks.

ELIGIBILITY:
Inclusion:

* Greater than 18 and less than 86 years of age;
* On stable medication regimen

  o Full-tolerated doses of 3 or more anti-hypertensive medications of different classes, one of which must be a diuretic (with no changes for a minimum of two months prior to screening) that is expected to be maintained without changes for at least 3 months.
* Office systolic blood pressure (SBP) of greater than 160 mmHg based on an average of 3 blood pressure readings measured at both initial screening visit
* The individual agrees to have all study procedures performed
* Willing to provide written consent
* Females with childbearing potential must not be pregnant.

Exclusion

* eGFR of < 45 mL/min/1.73m2, using the MDRD calculation.
* More than one in-patient hospitalization for an anti-hypertensive crisis within the year.
* More than one episode(s) of orthostatic hypotension (reduction of SBP of ≥ 20 mmHg of diastolic blood pressure (DBP) of ≥ 10 mmHg within 3 minutes of standing).
* History of myocardial infarction (MI), unstable angina pectoris, syncope or a cardiovascular accident within 6 months of screening period
* Clinically significant atrioventricular (AV) conduction disturbances and/or arrhythmias (e.g. 2nd or 3rd degree AV block);
* Current of past history of heart failure (≤40% left ventricular ejection fraction (EF).
* Major of psychotropic agents and antidepressants.
* Use of nonsteroidal anti-inflammatory drug (NSAIDs)
* Known hypersensitivity or contraindication to Minocycline or other tetracycline.
* Smoking
* Concurrent severe disease (such as neoplasm or HIV positive or AIDS).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-30 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Reduction of ambulatory blood pressure | Change in baseline to week 54
  Change in systolic blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Carl Pepine, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health Cardiovascular Clinic, Gainesville, Florida, United States